CLINICAL TRIAL: NCT05983003
Title: Research on Identifying and Treatment Prognosis of Chronic Rhinosinusitis Based on Image and Sequencing Data
Status: Completed | Type: Observational
Sponsor: Zheng Liu (Other)
Collaborators: Wuhan Central Hospital (Other); First Affiliated Hospital of Zhongshan Medical University (Other); Clifford Hospital, Guangzhou, China (Other); The First Affiliated Hospital of Zhengzhou University (Other); Shanxi Bethune Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Xiangyang Central Hospital (Other); Longgang District People's Hospital of Shenzhen (Other); Wuhan Integrated Traditional Chinese and Western Medicine Hospital (Other); Wuhan Third Hospital (Other); Yangxin Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Zheng Liu, Professor of Otolaryngology-Head & Neck Surgery Vice Director Department of ENT Tongji Hospital Tongji Medical College Huazhong University of Science and Technology Affiliation: Huazhong University of Science and Technology, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: ENT-Radiology-01
Record Dates: First submitted 2023-07-30; First posted 2023-08-09 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Chronic Sinusitis; Radiology; Pathology; Surgery; Progression
Keywords: Chronic Sinusitis; Radiology; Progression
MeSH Terms: conditions — Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — For patients with chronic sinusitis undergoing surgical treatment, nasal polyps or ethmoid sinus lesion mucosa will be collected during the operation. For the control group, mucosa will be taken from patients undergoing surgery for nasal septum deviation or nasal sinus trauma, and normal ethmoid sinus mucosa or inferior turbinate tissue will be collected during the operation. The collected tissue specimens will be divided into two parts, with one part being fixed in 4% paraformaldehyde and the other part stored at -80°C.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Following the efficacy assessment method outlined in the 2020 EPOS guidelines, the treatment outcomes of chronic sinusitis are categorized as "controlled" or "uncontrolled." Clinical reference evaluation criteria include: nasal congestion, rhinorrhea, facial pain, reduced sense of smell, sleep disturbances, the need for ongoing medication maintenance and the abnormal nasal endoscopy findings, .If there are no three or more symptoms rated five or higher, the patient's chronic sinusitis is considered controlled.
  Interventions: Procedure: endoscopic sinus surgery
- Uncontrol: Following the efficacy assessment method outlined in the 2020 EPOS guidelines, the treatment outcomes of chronic sinusitis are categorized as "controlled" or "uncontrolled." Clinical reference evaluation criteria include: nasal congestion, rhinorrhea, facial pain, reduced sense of smell, sleep disturbances, the need for ongoing medication maintenance and the abnormal nasal endoscopy findings, . The classification is based on the number and severity of these symptoms,and patients with three or more symptoms rated five or higher are considered to have uncontrolled disease
  Interventions: Procedure: endoscopic sinus surgery

INTERVENTIONS:
Procedure: endoscopic sinus surgery — Open the sinus ostium, improve anatomical issues and remove the diseased tissue.
  Other Names: ESS

SUMMARY:
This project focuses on researching chronic rhinosinusitis in patients, employing image processing techniques and molecular biology methods to jointly determine the research objectives:

1. Investigating heterogeneity.
2. Developing an intelligent assessment model.
3. Creating a visual tool for diagnosis and prognosis.

DETAILED DESCRIPTION:
1. Investigating the heterogeneity of chronic rhinosinusitis: the project will utilize high-throughput information from various sources such as radiology, pathology, and proteomics to gain insights into the multi-dimensional and big data aspects of chronic rhinosinusitis. By analyzing this data, the study aims to identify and understand the different subtypes with more precise and personalized treatment approaches.
2. Developing an intelligent assessment model: using artificial intelligence algorithms, the project will analyze multi-omics data gathered from the research. The goal is to establish an intelligent assessment model that can accurately interpret the data and provide valuable insights into chronic rhinosinusitis.
3. Creating a visual tool for diagnosis and prognosis: the project seeks to integrate multi-omics information to establish an AI model for typing and prognostic prediction. By achieving these research objectives, this project aspires to enhance the understanding of chronic rhinosinusitis and contribute to the development of more precise, personalized, and effective treatment strategies for patients suffering from this condition.

ELIGIBILITY:
Inclusion Criteria:

1. oral glucocorticoid, and intranasal steroid spray and steroid irrigation treatment were discontinued at least 3 months and 1 month before surgery, respectively;
2. without acute asthma episode or acute upper airway infection within 1 month before surgery;
3. not under allergen immunotherapy or biologic treatment.

Exclusion Criteria:

1. fungal sinusitis;
2. antrochoanal polyps;
3. cystic fibrosis, vasculitis, primary ciliary dyskinesia, or immunodeficiency;
4. odontogenic maxillary sinusitis;
5. patients with history of craniocerebral trauma or sinonasal tumours.
6. insufficient CT quality (e.g., metal artifacts, motion artifacts, and lack of intact CT scan of sinuses);
7. slice thickness more than 2.5 mm.
8. women must not be pregnant, or breast-feeding;
9. patients with serious metabolic, cardiovascular, autoimmune, neurology, blood, digestive, cerebrovascular, or respiratory system disease, or any disease interfering with the evaluation of results or affecting subjects safety are excluded, such as glaucoma and tuberculosis;
10. patients with emotional or mental problems are excluded;
11. patients unsuitable for inclusion based on judgement of researchers are excluded;

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic rhinosinusitis (CRS) was diagnosed according to the international guideline European position paper on rhinosinusitis and nasal polyps (EPOS) 2020. All the patients had ongoing symptoms after initial attempts on medical treatments and underwent endoscopic sinus surgery.
Sampling Method: Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2024-04 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline at months 12 in visual analogue scale (VAS) after surgical intervention | 12month
  The VAS for rhinosinusitis was used to evaluate the total disease severity. The participants were asked to indicate on a 10 centimeters (cm) VAS the answer to the question, "How troublesome are your symptoms of your rhinosinusitis?" The range of the VAS was from 0 (not troublesome) to 10 (worse thinkable troublesome) of troublesome, where higher score indicated worse thinkable troublesome.

SECONDARY OUTCOMES:
Change from baseline at months 1, 3, 6 and 12 in 22-item sino-nasaloutcome test (SNOT-22) scores after surgical intervention | 1month, 3month, 6month, 12month
  The SNOT-22 is a validated questionnaire that was used to assess the impact of chronic rhinosinusitis on health-related quality of life (HRQoL). It is a 22 item questionnaire with each item assigned a score ranging from 0 (no problem) to 5 (problem as bad as it can be). The total score may range from 0 (no disease) to 110 (worst disease), lower scores representing better health related quality of life.
Revision surgery rate | 12month
  The rate of reoperation in each group after surgery
Symptom duration | 1month, 3month, 6month, 12month
  The time of duration of major symptoms of postoperative patients
Change from baseline at months 1, 3, 6 and 12 in nasal endoscopic score after surgical intervention | 1month, 3month, 6month, 12month
  Endoscopic result is scored according to Lund-Kennedy system, with the assessment of nasal polyp (NP), edema, nasal discharge, scarring and crusting. Items including edema, nasal discharge, scarring and crusting score 0 for no problem, 1 for mild abnormalities and 2 for severe abnormalities. NP score is graded and based on NP size recorded as the sum of the right and left nostril scores with a range of 0-8; higher scores indicate worse status. Individual score ranges from 0 (no polyps) to 4 (large polyps causing almost complete congestion/ obstruction of the inferior meatus) within each nostril.
Postoperative medication | 1month, 3month, 6month, 12month
  The duration and dose of postoperative medication needed to relieve symptoms

OTHER OUTCOMES:
Changes from baseline at months 1, 3, 6 and 12 in molecular indices of nasal lavage fluid by Bio-plex | 1month, 3month, 6month, 12month
  Investigate the change of inflammation molecular biomarkers using sample of nasal lavage fluid or mucosal lesion tissue. Biomarkers including interleukin 9, monocyte chemoattractant protein-1, macrophage inflammatory protein-1β, macrophage inflammatory protein-1α and chemokine (C-C motif ) ligand 17 in nasal lavage fluid by Bio-plex (Bio-Rad, Hercules, CA, USA) at months 1, 3, 6 and 12 were detected to compare the changes of molecular indices relative to baseline.
Changes from baseline at months 1, 3, 6 and 12 in molecular indices of nasal lavage fluid by ELISA | 1month, 3month, 6month, 12month
  Investigate the change of inflammation molecular biomarkers using sample of nasal lavage fluid or mucosal lesion tissue. Biomarkers including Immunoglobulin (Ig) E in nasal lavage fluid by enzyme linked immunosorbent assay (ELISA) at months 1, 3, 6 and 12 were detected to compare the changes of molecular indices relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Liu, Doctor, Principal Investigator — Huazhong University of Science and Techology
Locations (1):
- Department of ENT, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fokkens WJ, Lund VJ, Hopkins C, Hellings PW, Kern R, Reitsma S, Toppila-Salmi S, Bernal-Sprekelsen M, Mullol J, Alobid I, Terezinha Anselmo-Lima W, Bachert C, Baroody F, von Buchwald C, Cervin A, Cohen N, Constantinidis J, De Gabory L, Desrosiers M, Diamant Z, Douglas RG, Gevaert PH, Hafner A, Harvey RJ, Joos GF, Kalogjera L, Knill A, Kocks JH, Landis BN, Limpens J, Lebeer S, Lourenco O, Meco C, Matricardi PM, O'Mahony L, Philpott CM, Ryan D, Schlosser R, Senior B, Smith TL, Teeling T, Tomazic PV, Wang DY, Wang D, Zhang L, Agius AM, Ahlstrom-Emanuelsson C, Alabri R, Albu S, Alhabash S, Aleksic A, Aloulah M, Al-Qudah M, Alsaleh S, Baban MA, Baudoin T, Balvers T, Battaglia P, Bedoya JD, Beule A, Bofares KM, Braverman I, Brozek-Madry E, Richard B, Callejas C, Carrie S, Caulley L, Chussi D, de Corso E, Coste A, El Hadi U, Elfarouk A, Eloy PH, Farrokhi S, Felisati G, Ferrari MD, Fishchuk R, Grayson W, Goncalves PM, Grdinic B, Grgic V, Hamizan AW, Heinichen JV, Husain S, Ping TI, Ivaska J, Jakimovska F, Jovancevic L, Kakande E, Kamel R, Karpischenko S, Kariyawasam HH, Kawauchi H, Kjeldsen A, Klimek L, Krzeski A, Kopacheva Barsova G, Kim SW, Lal D, Letort JJ, Lopatin A, Mahdjoubi A, Mesbahi A, Netkovski J, Nyenbue Tshipukane D, Obando-Valverde A, Okano M, Onerci M, Ong YK, Orlandi R, Otori N, Ouennoughy K, Ozkan M, Peric A, Plzak J, Prokopakis E, Prepageran N, Psaltis A, Pugin B, Raftopulos M, Rombaux P, Riechelmann H, Sahtout S, Sarafoleanu CC, Searyoh K, Rhee CS, Shi J, Shkoukani M, Shukuryan AK, Sicak M, Smyth D, Sindvongs K, Soklic Kosak T, Stjarne P, Sutikno B, Steinsvag S, Tantilipikorn P, Thanaviratananich S, Tran T, Urbancic J, Valiulius A, Vasquez de Aparicio C, Vicheva D, Virkkula PM, Vicente G, Voegels R, Wagenmann MM, Wardani RS, Welge-Lussen A, Witterick I, Wright E, Zabolotniy D, Zsolt B, Zwetsloot CP. European Position Paper on Rhinosinusitis and Nasal Polyps 2020. Rhinology. 2020 Feb 20;58(Suppl S29):1-464. doi: 10.4193/Rhin20.600. PMID 32077450
- [Result] Hu Y, Cao PP, Liang GT, Cui YH, Liu Z. Diagnostic significance of blood eosinophil count in eosinophilic chronic rhinosinusitis with nasal polyps in Chinese adults. Laryngoscope. 2012 Mar;122(3):498-503. doi: 10.1002/lary.22507. Epub 2012 Jan 17. PMID 22252861